CLINICAL TRIAL: NCT03266445
Title: A Prospective, Randomized Trial of the Effect of Standard of Care Reduced Dose Versus Full Dose Buprenorphine/Naloxone in the Perioperative Period on Pain Control and Post Operative Opioid Use Disorder Symptoms
Brief Title: Effect of Buprenorphine/Naloxone Continuation on Pain Control and Opioid Use
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aurora Naa-Afoley Quaye, Instructor M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P001425
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Opioid-use Disorder; Pain, Acute; Surgery
Keywords: relapse; buprenorphine/naloxone; opioids; narcotics; post-surgical pain
MeSH Terms: conditions — Opioid-Related Disorders; Acute Pain; Recurrence; Pain, Postoperative | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to be maintained on their daily dose of buprenorphine/naloxone or to have their buprenorphine/naloxone reduced to 8mg prior to surgery. Each group will have identical perioperative treatment plans. Primary outcome measured is pain scores following surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FULL-BUPRENORPHINE (Active Comparator): Participants will be randomly assigned to be maintained on their daily dose of buprenorphine/naloxone
  Interventions: Drug: buprenorphine/naloxone
- LOW-BUPRENORPHINE (control) (No Intervention): Participants will be randomly assigned to have their daily dose of buprenorphine/naloxone reduced to 8mg on the day of surgery

INTERVENTIONS:
Drug: buprenorphine/naloxone — The intervention will be to either continue taking buprenorphine/naloxone or to have the medication reduced perioperatively.
  Other Names: Reduction vs Continuation
  Arms: FULL-BUPRENORPHINE

SUMMARY:
The aim of this study is to determine the effect of continuation of buprenorphine/naloxone in patients with history of Opioid Use Disorder (OUD) scheduled for surgery compared to reduced dose buprenorphine/naloxone prior to surgery on pain scores, opioid consumption, depressive symptoms and severity of substance use dependence- including record of problematic use of any non-prescribed opioids, alcohol and illicit narcotics.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) is characterized by non-remitting cycles of remission and opioid abuse relapse. It is associated with a high rate of psychiatric and physical co-morbidity when left untreated. Buprenorphine and buprenorphine/naloxone are effective opioid maintenance therapy (OMT) for OUD, however, treatment of acute post-surgical pain in patients taking buprenorphine is perceived to be challenging. Although not substantiated in clinical studies, the combination of high receptor binding affinity, long half-life, and partial mu opioid receptor agonism with buprenorphine/naloxone are thought to inhibit the analgesic actions of full mu opioid receptor agonists, potentially making standard postoperative pain control strategies less effective. There is no evidence based standard of care for optimal acute pain management strategies for patients taking buprenorphine and most recommendations are based upon provider opinion- occasionally conflicting along specialty lines. Some providers, mainly consisting of surgeons and anesthesiologists, recommend that buprenorphine should be discontinued at least 72 hours prior to elective surgery and replaced with low dose opioid agonists, in the interim. Other providers, mainly comprising of psychiatrists, contend that these patients should be maintained on buprenorphine throughout the peri-operative period at either a full or reduced dose to prevent an indeterminate risk of substance abuse relapse that can occur as consequence to the abrupt termination buprenorphine in the highly stressful surgical period. This study aims to inform this important unresolved question in the clinical care of this growing population. The investigators seek to determine the effectiveness of managing postoperative pain in patients with OUD where buprenorphine/naloxone is continued perioperatively compared to patients where buprenorphine/naloxone is reduced to a lower dose. Longitudinally, the investigators also intend to determine if there is a difference in substance abuse relapse in patients where buprenorphine/naloxone is continued vs. held by using self assessments and communication with the participant's buprenorphine provider.

ELIGIBILITY:
Inclusion Criteria:

* currently taking buprenorphine or buprenorphine/naloxone daily for treatment of opioid use disorder by DSM-V criteria
* on buprenorphine or buprenorphine/naloxone dose of greater than 8mg for at least 30 days
* ASA health class I-III

Exclusion Criteria:

* Unable to consent to the study
* Significant pulmonary or cardiac disease
* Renal insufficiency with a glomerular filtration rate less than 30ml/min
* Liver cirrhosis with a Model for End-Stage Liver Disease (MELD) score of greater than 25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-10-05 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-26 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain scores | 24 hours after surgery
  Level of pain on a Visual Analog Scale of 0-100 (0=no pain; 100=worst pain imaginable) This scale will be used to quantify the varying degrees of pain or discomfort experienced by the participant.

SECONDARY OUTCOMES:
Postoperative opioid consumption | 24 hours, 48 hours and 72 hours after surgery
  Amount of opioids needed for pain control postoperatively
Post-operative pain scores | 48 hours, 72 hours after surgery
  Level of pain on Visual Analog Scale 0-100 (0= no pain 100= worst pain imaginable) We will compare the results of the 48 and 72 hour time-points with the 24 hour time-point.
Presence, severity of substance abuse | 1 month after surgery
  Participants will complete questionnaires to identify the presence and severity of substance abuse.These values will be compared with baseline values obtained preoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Quaye, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to researchers involved in the study. All data will be collected and stored securely using the Redcap system to preserve privacy and confidentiality. Information regarding substance abuse history, including illicit narcotic use, will remain confidential and personal identifiers will be removed during data storage. Only members of the research team will have access to the data that participants have consented to provide. Participants will be informed that they have the right to not answer any question that makes them feel uncomfortable.

REFERENCES:
- [Background] McLellan AT, Lewis DC, O'Brien CP, Kleber HD. Drug dependence, a chronic medical illness: implications for treatment, insurance, and outcomes evaluation. JAMA. 2000 Oct 4;284(13):1689-95. doi: 10.1001/jama.284.13.1689. PMID 11015800
- [Background] Scott CK, Dennis ML, Laudet A, Funk RR, Simeone RS. Surviving drug addiction: the effect of treatment and abstinence on mortality. Am J Public Health. 2011 Apr;101(4):737-44. doi: 10.2105/AJPH.2010.197038. Epub 2011 Feb 17. PMID 21330586
- [Background] Degenhardt L, Bucello C, Mathers B, Briegleb C, Ali H, Hickman M, McLaren J. Mortality among regular or dependent users of heroin and other opioids: a systematic review and meta-analysis of cohort studies. Addiction. 2011 Jan;106(1):32-51. doi: 10.1111/j.1360-0443.2010.03140.x. Epub 2010 Nov 4. PMID 21054613
- [Background] Schuckit MA. Treatment of Opioid-Use Disorders. N Engl J Med. 2016 Jul 28;375(4):357-68. doi: 10.1056/NEJMra1604339. No abstract available. PMID 27464203
- [Background] Gordon AJ, Lo-Ciganic WH, Cochran G, Gellad WF, Cathers T, Kelley D, Donohue JM. Patterns and Quality of Buprenorphine Opioid Agonist Treatment in a Large Medicaid Program. J Addict Med. 2015 Nov-Dec;9(6):470-7. doi: 10.1097/ADM.0000000000000164. PMID 26517324
- [Background] Roberts DM, Meyer-Witting M. High-dose buprenorphine: perioperative precautions and management strategies. Anaesth Intensive Care. 2005 Feb;33(1):17-25. doi: 10.1177/0310057X0503300104. PMID 15957687
- [Background] Bryson EO. The perioperative management of patients maintained on medications used to manage opioid addiction. Curr Opin Anaesthesiol. 2014 Jun;27(3):359-64. doi: 10.1097/ACO.0000000000000052. PMID 24500338
- [Background] McCormick Z, Chu SK, Chang-Chien GC, Joseph P. Acute pain control challenges with buprenorphine/naloxone therapy in a patient with compartment syndrome secondary to McArdle's disease: a case report and review. Pain Med. 2013 Aug;14(8):1187-91. doi: 10.1111/pme.12135. Epub 2013 May 3. PMID 23647815
- [Background] Huang A, Katznelson R, de Perrot M, Clarke H. Perioperative management of a patient undergoing Clagett window closure stabilized on Suboxone(R) for chronic pain: a case report. Can J Anaesth. 2014 Sep;61(9):826-31. doi: 10.1007/s12630-014-0193-y. Epub 2014 Jul 2. PMID 24985936
- [Background] Kornfeld H, Manfredi L. Effectiveness of full agonist opioids in patients stabilized on buprenorphine undergoing major surgery: a case series. Am J Ther. 2010 Sep-Oct;17(5):523-8. doi: 10.1097/MJT.0b013e3181be0804. PMID 19918165
- [Background] Macintyre PE, Russell RA, Usher KA, Gaughwin M, Huxtable CA. Pain relief and opioid requirements in the first 24 hours after surgery in patients taking buprenorphine and methadone opioid substitution therapy. Anaesth Intensive Care. 2013 Mar;41(2):222-30. doi: 10.1177/0310057X1304100212. PMID 23530789
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Background] Wilkinson KM, Krige A, Brearley SG, Lane S, Scott M, Gordon AC, Carlson GL. Thoracic Epidural analgesia versus Rectus Sheath Catheters for open midline incisions in major abdominal surgery within an enhanced recovery programme (TERSC): study protocol for a randomised controlled trial. Trials. 2014 Oct 21;15:400. doi: 10.1186/1745-6215-15-400. PMID 25336055
- See also: Center for Behavioral Health Statistics and Quality. Behavioral health trends in the United States: Results from the 2014 National Survey on Drug Use and Health. 2015. HHS Publication No. SMA 15-4927, NSDUH Series H-50. — https://www.samhsa.gov/data/sites/default/files/NSDUH-FRR1-2014/NSDUH-FRR1-2014.pdf